CLINICAL TRIAL: NCT06028503
Title: Effectiveness of a Community-Based Intervention of Acceptance and Commitment Therapy for Type 2 Diabetes Management in a Rural and Underserved Community
Brief Title: ACT Intervention for Type 2 Diabetes Management for Rural and Underserved Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sam Houston State University (Other)
Collaborators: Chelsea Ratcliff, Ph.D. (Unknown); Owen Kelly, Ph.D.,RNutr (Unknown); Oluwaseun Olaiya, DO (Unknown); Michael Griffin, Ph.D. (Unknown)
Responsible Party: Principal Investigator, Ryan J Marek, Ph.D., Assistant Professor of Clinical Psychology, Sam Houston State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2023-194
Record Dates: First submitted 2023-07-31; First posted 2023-09-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: his study will compare the efficacy of ACT+CGM+LE to CGM+LE, or LE alone, on hemoglobin HbA1c in 60 people with T2D recruited from a rural population.
Who Masked: Participant
Masking Description: The RC will have a shuffled stack of envelopes with a group assignment in each. As participants meet inclusion into the study, their information, including Study ID, will be placed in one of the shuffled envelopes. The envelope will be placed in another envelope and sealed. Once approximately 10 participants are randomized to each group, the RC will contact all participants who have been randomized to share the date and time of the intervention and ask them to complete the 30-minute baseline surveys comprised of self-report measures (located in measures section) that they will receive by email. If recruitment slows down, we will do the randomization once 5 participants express interest in the study. The RC will then send a unique Qualtrics link to each participant (to prevent participants from needing to enter identifying information on the survey). The baseline self-report survey is described below in the Measures section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acceptance and Commitment Therapy + Continuous Glucose Monitoring + Lifestyle Education (ACT+CGM+LE) (Experimental): Participants assigned to ACT+CGM+LE will have both of the above modules in addition to three ACT modules based on Gregg et al.8 and traditional ACT therapy19. Two facilitators will lead the ACT sessions: Dr. Marek or Dr. Ratcliff and one trained doctoral-level clinical psychology student under their direct supervision (i.e., one licensed provider paired with a student). We will run all sessions in a group format. Participants will be given breaks between modules and one long lunch break.
  Interventions: Behavioral: Acceptance and Commitment Therapy; Device: Abbott FreeStyle® Libre® 3; Other: Generic Education
- Continuous Glucose Monitoring + Lifestyle Education (CGM+LE) (Experimental): Participants assigned to CGM+LE will attend the group LE workshop. CGM training will occur after the 5 hour lifestyle education delineated above (same content, but less informal discussion). This will include training on using blood glucose monitoring devices, setting up the App on the smartphone (including activating the hypoglycemic alarm) and how to apply the glucose sensors on the arm. If a sensor does fall off a participant, a member of the study team will provide a spare sensor to the participant. The glucose range for participants will be set at between 70 and 140 mg/dL, unless the study physician (Dr. Olaiya) determines otherwise. The CGM device will allow us to calculate the percentage of 'time in range' per day, peak glucose, nocturnal glucose and number of hypoglycemic events. The CGM training will be managed by Dr. Olaiya and/or Dr. Kelly, and a medical/dietetic students.
  Interventions: Device: Abbott FreeStyle® Libre® 3; Other: Generic Education
- Lifestyle Education (LE) (Active Comparator): Participants will be given information about how lifestyle choices, including daily dietary choices, affect blood sugar for people with T2D, and best practices related to checking blood sugar and carbohydrate counting if participants are on insulin therapy.
  Interventions: Other: Generic Education

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Approximately 3 hours of ACT will be administered based on Gregg et al.;s (2007) protocol:
  1. What is ACT?
  2. Coping and Stress Management
  3. Acceptance and Action
  Arms: Acceptance and Commitment Therapy + Continuous Glucose Monitoring + Lifestyle Education (ACT+CGM+LE)
Device: Abbott FreeStyle® Libre® 3 — The Abbott FreeStyle® Libre® 3 (FDA approved) consists of a single use disposable electrochemical sensing unit which is placed on the upper arm and an App for smart phones where the participant can view their glucose data, including their current glucose reading, their 'trend arrow' so participants can see how glucose is changing, and their glucose history. The FreeStyle system does not require user calibration. A sensor log will be maintained for accountability of all sensors received as well as used sensors (including the lot/serial number, expiration date, and the date). Sensors will be stored at manufacturers recommendations.
  Arms: Acceptance and Commitment Therapy + Continuous Glucose Monitoring + Lifestyle Education (ACT+CGM+LE); Continuous Glucose Monitoring + Lifestyle Education (CGM+LE)
Other: Generic Education — Participants will be given information about how lifestyle choices, including daily dietary choices, affect blood sugar for people with T2D, and best practices related to checking blood sugar and carbohydrate counting if participants are on insulin therapy. These sessions will also include education on diabetes nutrition guidelines and improving self-management through better food and lifestyle choices.

SUMMARY:
The purpose of this project is to examine the feasibility/acceptability of a one-day Acceptance and Commitment Therapy + Lifestyle Education group intervention paired with 12-weeks of Continuous Glucose Monitoring for patients with type 2 diabetes (T2D) living in rural communities. This study is being designed as a randomized control trial (RCT) comparing ACT+LE+CGM to LE+CGM to LE. The ultimate goal of this line of research is that a community-wide intervention of Acceptance and Commitment Therapy (ACT) with Continuous Glucose Monitoring (CGM) and Lifestyle Education (LE) will improve T2D outcomes in rural communities compared to CGM and LE, or LE alone. Our goal is to develop a scalable and sustainable program for diabetes management in rural areas that enables individual self-management and does not require extensive healthcare resources in an existing medical desert.

DETAILED DESCRIPTION:
ADA guidelines highlight the essential role of nutrition therapy and/or diabetes self-management education (DSME) programs in diabetes management. A recent NHANES analysis which included 2365 people with diabetes indicated that only 32% are considered in good control of diabetes (HbA1c 6.5-6.9%). In the rural community at higher risk of diabetes, conventional lifestyle intervention approaches to diabetes management (e.g., Look AHEAD) or prevention, are not sustainable as they are resource intense. In medical deserts such as rural areas, there is a need for alternative strategies. To add, a mechanism that can impact lack of behavioral adherence is experiential avoidance. Experiential avoidance describes avoiding or escaping behaviors that cause B. distress, anxiety, shame, guilt, pain, and others. Acceptance and Commitment Therapy (ACT) targets experiential avoidance, which many believe prevents engagement in health behavior change. ACT has demonstrated efficacy in numerous psychological and biomedical diseases, including depression and anxiety, migraines, chronic pain, inflammatory bowel disease, weight loss, and T2D. ACT helps patients to overcome avoidance of health behaviors by promoting acceptance of negative feelings and thoughts and by encouraging them to engage in behaviors that align well with their values. Although dietary data suggest people with diabetes may be making self-perceived positive dietary changes, experiential avoidance likely prohibits sustained food behavior change and better self-management.

The purpose of this project is to examine the feasibility/acceptability of a one-day Acceptance and Commitment Therapy + Lifestyle Education group intervention paired with 12-weeks of Continuous Glucose Monitoring for patients with type 2 diabetes (T2D) living in rural communities. This study is being designed as a randomized control trial (RCT) comparing ACT+LE+CGM to LE+CGM to LE. The ultimate goal of this line of research is that a community-wide intervention of Acceptance and Commitment Therapy (ACT) with Continuous Glucose Monitoring (CGM) and Lifestyle Education (LE) will improve T2D outcomes in rural communities compared to CGM and LE, or LE alone. Our goal is to develop a scalable and sustainable program for diabetes management in rural areas that enables individual self-management and does not require extensive healthcare resources in an existing medical desert.

Specific aims:

Aim 1: To implement and adapt (to include CGM monitoring) an abbreviated (one day session) ACT protocol for T2D8 that we can administer at the group level to rural individuals. By the end of the one-day workshop, participants should understand how to use acceptance skills (e.g., mindfulness, cognitive defusion from negative thoughts) to engage in committed action towards T2D management and adherence. Two clinical psychologists, with input from the multidisciplinary team, will adapt the protocol and participant worksheets from existing brief ACT interventions for T2D.

Aim 2: To conduct a pilot single-blind randomized control trial of an adapted ACT for T2D, in combination with CGM and LE, to evaluate the feasibility, acceptability and initial efficacy of this protocol at a among in rural individuals. Therefore, this study will compare the efficacy of ACT+CGM+LE to CGM+LE, or LE alone, on hemoglobin HbA1c in 60 people with T2D recruited from a rural population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed diabetes (self-reported) and with an HbA1c ≥ 6.0 (using point-of-care device)
2. at least 18 years of age or older
3. able to speak English
4. able to provide informed consent and participate in the study
5. reliable access to a personal smartphone device 6) zip code is associated with a rural area.

Exclusion Criteria:

1. Reported suicidal ideation at the initial visit
2. has evidence of acute psychosis that precludes informed consent
3. appears to be cognitively impaired to the extent that precludes informed consent
4. uses a heavy amount of alcohol or other substances
5. is deemed by the multidisciplinary study team has too medically complex for a more conservative treatment approach
6. has a pacemaker or other implanted electrical medical device
7. Pregnant (management of diabetes while pregnant may require additional medical oversight).
8. Under 18 years old (protocol was validated for adults)
9. Non-English-speaking individuals (protocol has not been translated and validated in other languages)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hemoglobin A1C | 1-year
  Our goal is to determine if CGM and ACT can change HbA1c 3 months after the intervention and to determine if those reductions can be sustained one year after the intervention.

SECONDARY OUTCOMES:
Body Mass Index | 1-year
  Body weight will be measured with the participant in light clothing without shoes. Body height will be measured to the nearest 0.1 cm without shoes using a calibrated stadiometer at screening only. Body weight and height will be used to calculate BMI (BMI = weight/height2 (kg/m2).
Body Composition | 1-Year
  Waist circumference will be measured at a level midway between the lower rib margin and iliac crest with the tape all around the body in a horizontal position, using a calibrated measuring tape.
Experiential Avoidance | 1-Year
  We will assess experiential avoidance with the Acceptance and Action Questionnaire - 2 (AAQ-2) - The AAQ-2 is a reliable and valid self-report measure of psychological flexibility and experiential avoidance.
Depression | 1-Year
  We will assess depression via the NIH Patient Report Outcomes Measures Information System (PROMIS) scale for depression. The NIH PROMIS measure for depression has eight items that reliably and validly assess the construct of depression.
Adherence | 1-Year
  We will administer the Diabetes Care Profile (DCP), which will assess our participants' frequency and adherence to regular blood sugar monitoring and their understanding of T2D.
Food Insecurity | 1-Year
  Food insecurity will be assessed using the USDA Economic Research Services U.S. Adult Food Security Survey Module. This validated survey tool has 10 items in a three-stage design with screeners. Screening keeps respondent burden to the minimum, which improves data reliability. This will allow us to explore if food insecurity impacts diabetes progression.
Health literacy | Baseline
  Health literacy will be measured using the Short Assessment of Health Literacy-English (SAHL-E) from the PhenX Toolkit. This includes 18 interviewer-administered items designed to assess the participants ability to read and understand common medical terms. This survey will be administered at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sam Houston State University College of Osteopathic Medicine, Conroe, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to place the data in an open data repository. We intend to reach out NIH's NIDDK's data repository to determine if they will let us store our data there to promote openness and transparency.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will adhere to all polices in the repository that will accept our data. Data will become available once primary outcome data is analyzed by the study team and reported or when the repository requires - whichever comes first.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT06028503/Prot_SAP_ICF_000.pdf